CLINICAL TRIAL: NCT04827498
Title: Myocardial Ischemia Without Obstructive Coronary Stenoses: A Prospective Observational Study With Invasive Coronary Pressure and Flow Measurements and Endothelial Function Test
Brief Title: Myocardial Ischemia Without Obstructive Coronary Stenoses
Status: Recruiting | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Responsible Party: Principal Investigator, Hernan D. Mejia-Renteria, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: 21/289-E
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Myocardial Ischemia; Non-Obstructive Coronary Atherosclerosis; Microvascular Coronary Artery Disease; Vasospastic Angina; Myocardial Bridging
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris, Variant; Myocardial Bridging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocardial ischemia without obstructive coronary stenosis
  Interventions: Diagnostic Test: Invasive coronary endothelium-dependent and non-endothelium-dependent physiological assessment

INTERVENTIONS:
Diagnostic Test: Invasive coronary endothelium-dependent and non-endothelium-dependent physiological assessment — Coronary hemodynamics and vessel anatomical measures obtained during adenosine and acetylcholine evaluation with a dedicated physiology wire

SUMMARY:
Coronary-related myocardial ischemia can result from obstructive epicardial stenosis or non-obstructive causes including coronary microcirculatory dysfunction and vasomotor disorders. This prospective study has been created in order to provide knowledge in the field of non-obstructive coronary artery disease.

DETAILED DESCRIPTION:
All-comer patients referred for coronary physiological assessment with pressure-flow measurements and acetylcholine endothelial function test, aimed to investigate different aspects of non-obstructive coronary artery disease, will be enrolled. Coronary hemodynamics during adenosine or acetylcholine evaluation will be measured either with a physiology wire equipped with pressure and temperature sensors (Abbott), or with a physiology wire equipped with pressure sensor and Doppler (Philips). Non-endothelium-dependent functional assessment will be performed with intravenous or intracoronary adenosine administration following the standard practice. Endothelium-dependent functional assessment will be performed with intracoronary acetylcholine bolus administration following the standard practice, which includes continuous 12-lead ECG monitorization. Microcirculatory dysfunction and vasomotor disorders will be diagnosed according to the criteria from the last European expert consensus on Ischaemia with Non-Obstructive Coronary Arteries (INOCA). Medical therapy will be adjusted on the basis of physiology study results and patients will be followed at 30 days, 1-, 2- and 5-years either at the outpatient clinic or by telephone contact. The Seattle Questionnaire of Angina will be applied during follow-up for obtaining an objective characterisation of the angina status.

OBJECTIVES OF THE STUDY:

* To investigate the coronary hemodynamics across the spectrum of coronary microcirculatory dysfunction.
* To investigate the coronary hemodynamics across the spectrum of vasomotor disorders.
* To investigate the impact of coronary microcirculatory dysfunction on clinical outcomes and patient symptoms at long-term follow-up.
* To investigate the impact of coronary vasomotor disorders on clinical outcomes and patient symptoms at long-term follow-up.
* To investigate the impact of a stratified medical therapy (guided by invasive physiology study) on patient symptoms.
* To investigate the role of microcirculatory dysfunction and vasomotor disorders in different settings of ischemic heart disease (i.e., recurrent angina despite successful percutaneous coronary intervention; myocardial infarction without obstructive coronary artery disease; left ventricular dysfunction (either systolic or diastolic) with or without heart failure).
* To develop new, alternative methods aimed to assess the coronary microcirculation.
* To investigate the role of myocardial bridging on myocardial ischemia generating mechanisms.
* To document safety of intracoronary testing in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent available.
* Age ≥ 18 years.
* Patient eligible for invasive physiological assessment with adenosine and / or acetylcholine.

Exclusion Criteria:

* Hemodynamic instability.
* Anticipated technical issues for physiology wire measurements.
* Culprit vessel of acute coronary syndrome
* Contraindications for adenosine administration.
* Contraindications for acetylcholine test.
* Reduced life expectancy (less than 1 year).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of patients with clinically indicated invasive physiological measures of coronary pressure and flow with adenosine and acetylcholine for the assessment of myocardial ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite outcome | Up to 5 years
  Incidence of a patient-oriented composite outcome, a composite of any death, nonfatal myocardial infarction, any ischemia-driven revascularization or hospitalization due to unstable angina pectoris
Vessel-oriented composite outcome | Up to 5 years
  Incidence of a vessel-oriented composite outcome, a composite of cardiac death, target-vessel related myocardial infarction or target-vessel revascularization
Patient symptoms burden | Up to 12 months
  Change in the Seattle questionnaire of angina scoring, associated to stratified medical treatment. Minimum is 0 and maximum is 100 and lower scores indicate worse outcome

SECONDARY OUTCOMES:
Cumulative incidence of any death | Up to 5 years
Cumulative incidence of cardiac death | Up to 5 years
Cumulative incidence of nonfatal myocardial infarction | Up to 5 years
Cumulative incidence of ischemia-driven revascularization | Up to 5 years
Safety of invasive comprehensive coronary functional testing with adenosine and acetylcholine | During procedure
  Adverse events / complications linked to invasive functional testing
Emergency room visit due to angina episode | Up to 5 years

OTHER OUTCOMES:
Resting and hyperemic mean aortic pressure (mmHg) | During procedure
  Measured with the coronary guiding catheter during physiology assessment under adenosine administration and acetylcholine provocation test
Resting and hyperemic mean intracoronary distal pressure (mmHg) | During procedure
  Measured with the coronary physiology wire under adenosine administration and acetylcholine provocation test
Resting and hyperemic mean coronary flow (mean transit time or cms/sec) | During procedure
  Measured with the coronary physiology wire under adenosine administration and acetylcholine provocation test
Resting and hyperemic coronary microcirculatory resistance (units) | During procedure
  Measured with the coronary physiology wire under adenosine administration and acetylcholine provocation test
Resting Pd/Pa (units) | During procedure
  Measured with the coronary physiology wire under resting conditions
Resting full cycle ratio (units) | During procedure
  Measured with the coronary physiology wire under resting conditions
Instantaneous wave-free ratio (units) | During procedure
  Measured with the coronary physiology wire under resting conditions
Fractional flow reserve (units) | During procedure
  Measured with the coronary physiology wire under hyperemia
Coronary flow reserve (units) | During procedure
  Measured with the coronary physiology wire under adenosine administration and acetylcholine provocation test
Resistive reserve ratio (units) | During procedure
  Measured with the coronary physiology wire under adenosine administration and acetylcholine provocation test
Location of vasospasm into the coronary vessel (proximal, mid or distal) | During procedure
  Detected under acetylcholine provocation test
Type of transient ischemic ECG changes (T wave inversion, ST depression, ST elevation) | During procedure
  Observed under acetylcholine provocation test
Change in diameter vessel (in percentage) | During procedure
  Measured with quantitative coronary angiography under acetylcholine and nitroglycerin intracoronary administration

CONTACTS AND LOCATIONS:
Overall Officials: Hernan Mejia-Renteria, MD, PhD, Principal Investigator — Department of Cardiology, Hospital Clinico San Carlos; Javier Escaned, MD, PhD, Principal Investigator — Department of Cardiology, Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study contemplates the possibility of sharing data with other researchers who have similar objectives. IPD to be shared includes demographic data, vessel characteristics, invasive coronary physiology data and outcome measures, appropriately anonymized.
Supporting Information: Study Protocol, CSR
Time Frame: Throughout the development of the study

REFERENCES:
- [Derived] Mejia-Renteria H, Shabbir A, Nunez-Gil IJ, Macaya F, Salinas P, Tirado-Conte G, Nombela-Franco L, Jimenez-Quevedo P, Gonzalo N, Fernandez-Ortiz A, Escaned J. Feasibility and Improved Diagnostic Yield of Intracoronary Adenosine to Assess Microvascular Dysfunction With Bolus Thermodilution. J Am Heart Assoc. 2024 Nov 19;13(22):e035404. doi: 10.1161/JAHA.124.035404. Epub 2024 Nov 7. PMID 39508144
- [Derived] Mejia-Renteria H, Wang L, Chipayo-Gonzales D, van de Hoef TP, Travieso A, Espejo C, Nunez-Gil IJ, Macaya F, Gonzalo N, Escaned J. Angiography-derived assessment of coronary microcirculatory resistance in patients with suspected myocardial ischaemia and non-obstructive coronary arteries. EuroIntervention. 2023 Apr 3;18(16):e1348-e1356. doi: 10.4244/EIJ-D-22-00579. PMID 36534493